CLINICAL TRIAL: NCT06629220
Title: Co-creation of Tools for Men With Suicidal Thoughts and/or Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0366
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Suicide Prevention; Suicidal Ideation; Suicidal Behaviour
Keywords: co-creation; participatory research; men; suicide prevention; suicidal ideation; male health
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Co-creation meetings (Other): All participants will be invited to participate in the co-creation meetings.
  Interventions: Other: Tools

INTERVENTIONS:
Other: Tools — In the co-creation meetings, developed tools will be presented. Participants will be asked to provide feedback and input to tailor these tools to the needs and preferences of men with suicidal thoughts/behavior.

SUMMARY:
The primary objective of this project is to co-create suicide prevention tools for men with suicidal thoughts ensuring these tools are supported by their future users. The researchers will organize up to 10 online or live co-creation meetings of maximum 2 hours each in which men (18 years or older) with a history of suicidal thoughts and/or behavior will help develop tools by providing their needs and feedback. Up to 30 men can participate.

DETAILED DESCRIPTION:
Approximately three out of four people who die by suicide are men. Suicide is a complex phenomenon, which cannot be explained by a single factor, but rather is a result of a variety of neuro-biological, psychological and social risk factors.

Considering the difference in suicide risk between men and women, researchers have tried to identify risk factors specific to men, which might contribute to the increased suicide risk. Differences in help-seeking behavior and received help have repeatedly been put forward as being one of these factors as men are less likely to seek help and have a higher drop-out rate once having started interventions.

A currently ongoing study (BUN: B6702024000090) focuses on mapping out these needs and barriers among adult men with suicidal thoughts and their healthcare providers.

The next step is to develop tools that meet the indicated needs and facilitate help-seeking and (continuous) help-receiving among men with suicidal thoughts and behavior. To develop these tools a co-creation process will be used, where men with a history of suicidal thoughts will be involved. Using the input of future users of tools is crucial. The investigators want to ensure that the developed tools are user-friendly for future users so that the barriers of using them remain as low as possible. The investigators want to do this by adapting the used language and layout to the preferences of our future users. In addition, the investigators want to ensure that the content in the tools is relevant and understandable for everyone. The investigators also aim to develop tools that appeal to a diverse group of users.

It is therefore crucial that the people who will use the tools are involved in their creation and design to suit their needs and use valuable experiential knowledge (Boyle, 2007; Hanlon et al., 2022; Watling et al., 2020). This is also called participatory co-creation. It means that men with a history of suicidal thoughts are at the center of the decision about how the tools should look. Additionally, experts on healthcare and masculinity, as well as international research literature will be consulted.

The primary objective of this project is to co-create suicide prevention tools for men with suicidal thoughts ensuring these tools are supported by their future users.

This will be done by maximum 10 live or online co-creation meetings with men (18 years or older) who experienced suicidal thoughts and/or behaviors in the past 3 years. The co-creation meetings will take place in groups with a maximum of 10 participants. Participants can participate in a minimum of 1 and a maximum of 10 co-creation meetings. The meetings will last a maximum of 2 hours. The co-creation meetings will be supervised and carried out by the Flemish Center of Expertise in Suicide prevention researchers.

If participants feel that participating in group is too much of a barrier, the investigators offer the possibility to have a one-on-one interview with the same content/questions. This exception allows us to gain information from all interested participants without excluding individuals due to their unwillingness or inability to participate in group. At the meeting, two researchers will be present and possibly people specialized in developing tools. The tools are developed in consultation with the developer, Flemish Center of Expertise in Suicide Prevention researchers, experts in the field and men with a history of suicidal thoughts.

After expressing interest to participate, participants will be contacted by telephone by one of the researchers to provide more information about the co-creation meetings and to answer any questions. During this phone call, a researcher (clinical psychologist) will evaluate the exclusion criteria. If the participant is interested in participating in the co-creation meetings and is eligible for participation, they will be asked to provide informed consent online. After providing consent, they will be asked to complete a short online background questionnaire on demographic characteristics because the researchers would like to ensure diversity and cultural and social aspects are considered in the tool development. The participants in the co-creation meetings must therefore be a representative group of the intended population. The participant will then receive the invitation to the meetings by email or text message.

ELIGIBILITY:
Inclusion Criteria:

* Men (≥ 18y/o)
* Experienced suicidal thoughts in the past three year

Exclusion Criteria:

* Limited comprehension
* Acute suicidality (as evaluated by a clinical psychologist of the research team)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified male participants can participate (based on gender and not sex)
Enrollment: 30 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Co-creation questions | From enrolment to end of co-creation sessions (10 sessions of 2 hours max over the course of the study)
  During the meetings, participants will be asked to provide feedback on developed tools and drafts (open questions). Here are some topics and questions the researchers will consider during the meetings:
  1. Current healthcare/tools usage
  2. Preferences and needs (this will be mainly based on the results of our previous study, BUN B6702024000090)
  3. Accessibility and usability of the tool
  4. Privacy and confidentiality
  5. Social support and sensitivity
  6. Help and professional support
  7. Continuity and long-term implementation
  8. Feedback on prototypes of the tool
  9. Feedback on final version of the tool

OTHER OUTCOMES:
Socio-demographic characteristics: gender | Baseline. Completing the entire 'socio-demographic characteristics questionnaire' will take about 5 minutes
  gender [male, female, non-binary, other]
Socio-demographic characteristics: age | Baseline. Completing the entire 'socio-demographic characteristics questionnaire' will take about 5 minutes
  age [open]
Socio-demographic characteristics: history of suicidal ideation | Baseline. Completing the entire 'socio-demographic characteristics questionnaire' will take about 5 minutes
  previous suicidal thoughts [never; more than 3 years ago, 1-3 years ago, in the past year]
Socio-demographic characteristics: education level | Baseline. Completing the entire 'socio-demographic characteristics questionnaire' will take about 5 minutes
  education [no degree, primary education, secondary education, higher education non-university, higher education university]
Socio-demographic characteristics: employment status | Baseline. Completing the entire 'socio-demographic characteristics questionnaire' will take about 5 minutes
  employment status [student, mainly employed, mainly self-employed, mainly houseman; looking for work, incapacitated, retired]
Socio-demographic characteristics: sexual orientation | Baseline. Completing the entire 'socio-demographic characteristics questionnaire' will take about 5 minutes
  sexual orientation [heterosexual, homosexual, bisexual, asexual, other, prefer not to say, dont know]
Socio-demographic characteristics: relationship status | Baseline. Completing the entire 'socio-demographic characteristics questionnaire' will take about 5 minutes
  relationship status [single, in relationship, married/cohabitant, separated, divorced, widowed]
Socio-demographic characteristics: living situation | Baseline. Completing the entire 'socio-demographic characteristics questionnaire' will take about 5 minutes
  living situation [alone, with partner, with children, with parents, with others, other - multiple options possible]
Socio-demographic characteristics: cultural background | Baseline. Completing the entire 'socio-demographic characteristics questionnaire' will take about 5 minutes
  cultural background [Belgian background, Western migration background, non-Western migration background, other]

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyle, E. (2007),
- [Background] Hanlon CA, McIlroy D, Poole H, Chopra J, Saini P. Evaluating the role and effectiveness of co-produced community-based mental health interventions that aim to reduce suicide among adults: A systematic review. Health Expect. 2023 Feb;26(1):64-86. doi: 10.1111/hex.13661. Epub 2022 Nov 14. PMID 36377305
- [Background] Watling D, Preece M, Hawgood J, Bloomfield S, Kolves K. Developing an Intervention for Suicide Prevention: A Rapid Review of Lived Experience Involvement. Arch Suicide Res. 2022 Apr-Jun;26(2):465-480. doi: 10.1080/13811118.2020.1833799. Epub 2020 Oct 18. PMID 33073734